CLINICAL TRIAL: NCT07326397
Title: Comparative Evaluation of Intrathecal Dexmedetomidine and Magnesium Sulphate as Adjuvants to 0.5% Hyperbaric Bupivacaine for Spinal Anesthesia in Patients Undergoing Dynamic Hip Screw (DHS) Fixation: A Randomized Clinical Study
Brief Title: Comparison Between Intrathecal Magnesium Sulphate & Dexmedetomidine in DHS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shehab Fathy Ahmed Osman, Resident doctor at Assiut University Hospital, Assiut, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Intrathecal Mgso4& Dex. In DHS
Record Dates: First submitted 2025-11-19; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Effects of Dexmedetomidine & Magnesium Sulphate on Patients Undergoing DHS
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Dexmedetomidine) (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Group M (Magnesium Sulphate) (Active Comparator)
  Interventions: Drug: Magnesium Sulphate

INTERVENTIONS:
Drug: Dexmedetomidine — 2.5 mL 0.5% hyperbaric bupivacaine + 5 µg dexmedetomidine (0.5 mL), total volume 3 mL
  Arms: Group D (Dexmedetomidine)
Drug: Magnesium Sulphate — 2.5 mL 0.5% hyperbaric bupivacaine + 50 mg magnesium sulphate (0.5 mL), total volume 3 mL
  Arms: Group M (Magnesium Sulphate)

SUMMARY:
To compare the efficacy and safety of intrathecal dexmedetomidine and magnesium sulphate as adjuvants to 0.5% hyperbaric bupivacaine in patients undergoing elective DHS fixation, focusing on onset and duration of sensory and motor block, hemodynamic stability, and quality of postoperative analgesia.

DETAILED DESCRIPTION:
Spinal anesthesia is a preferred technique for lower limb orthopedic surgeries due to its rapid onset, reliable sensory and motor blockade, and minimal systemic side effects. Hyperbaric bupivacaine 0.5% is commonly used; however, its duration may be insufficient for prolonged procedures or postoperative analgesia. To enhance and prolong anesthesia and analgesia, various intrathecal adjuvants have been investigated.

Dexmedetomidine, a selective α2-adrenergic agonist, has shown promise in improving the quality and duration of spinal anesthesia by providing prolonged sensory and motor blockade, stable hemodynamics, and enhanced postoperative analgesia. Similarly, magnesium sulphate, an NMDA receptor antagonist, exerts antinociceptive effects by modulating calcium influx in nerve cells, potentially prolonging analgesia without significant motor blockade.

Dynamic hip screw (DHS) fixation is a common surgical intervention for intertrochanteric femur fractures, particularly in elderly patients. These procedures demand reliable intraoperative anesthesia and effective postoperative pain control to facilitate early mobilization and reduce complications.

Despite individual studies evaluating these agents, direct comparisons between intrathecal dexmedetomidine and magnesium sulphate as adjuvants to bupivacaine in DHS fixation remain limited. This study aims to compare their efficacy and safety in enhancing spinal anesthesia, thereby optimizing perioperative care in patients undergoing elective DHS fixation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 year
* ASA Physical Status I or II
* Scheduled for elective DHS fixation under spinal anesthesia
* Written informed consent provided
* Patients of both sex are included in the study.

Exclusion Criteria:

* Patient refusal
* Allergy to study drugs
* Local infection at injection site
* Neurological or psychiatric illness
* Coagulopathy
* Chronic opioid or sedative use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Highest Dermatome Level of Sensory Block | 24 hours after intervention
  Sensory block level assessed using a pinprick test and recorded as the highest dermatome level with loss of sensation.
Duration of postoperative analgesia | 24 hours after intervention
  The outcome is Measured by Vas Score to assess pain intensity. It consists of a numeric version of the visual analogue scale. It is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible. This scale can be administered verbally. Vas score for 24 h will be assessed at 0., 1, 12 and 24 h postoperatively and will be recorded.
Degree of Motor Block | 24 hours after intervention
  Motor block assessed using the Modified Bromage Scale (0-3), where higher scores indicate greater motor block.

SECONDARY OUTCOMES:
Heart Rate | 24 hours after intervention
  Heart rate measured in beats per minute (bpm)
Incidence of Adverse Effects | 24 hours after Intervention
  Bradycardia Hypotension Nausea Vomiting Sedation (Assessed By Ramsay Sedation Scale (RSS) ) Shivering Respiratory depression Delayed motor block Flushing Warm sensation Headache Pruritus Urinary retention Neurological complications (e.g., transient paresthesia)
Mean Arterial Pressure | 24 hours after intervention
  Mean arterial pressure measured in mmHg
Oxygen Saturation | 24 hours after intervention
  Peripheral oxygen saturation measured by pulse oximetry by percentage